CLINICAL TRIAL: NCT06679777
Title: Swedish CArdioPulmonary bioImage Study 2
Acronym: SCAPIS2
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Lund University (Other); Uppsala University (Other); Umeå University (Other); Linkoeping University (Other Government); Göteborg University (Other)
Responsible Party: Principal Investigator, Tomas Jernberg, Professor, Karolinska Institutet
Other Study IDs: 2024-01
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Diseases; Lung Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the Swedish CArdioPulmonary bioImage Study (SCAPIS 1), 30,154 randomly selected men and women, aged 50-64 years, were recruited from six areas in Sweden during 2013-2018. The study population was investigated with CCTA, ultrasound carotids, physical examination, questionnaires, accelerometry, ECG, spirometry, and biochemical markers. The aim was to obtain new information relevant to the identification and treatment of individuals with cardiopulmonary and metabolic diseases and to optimize the possibilities for studying disease mechanisms.

In SCAPIS-2, half of the individuals (n≈15,000) included in SCAPIS 1, will be re-examined 2024-2025 with the same investigations as during 2013-2018 except for ultrasound of the carotids.

DETAILED DESCRIPTION:
The overall aim of SCAPIS is to improve prediction and prevention of cardiovascular and lung disease in the general population by identifying novel risk markers. This is also the purpose of SCAPIS 2, which further aims to gain important insights into risk factors and longitudinal development of heart, vascular and lung diseases such as atherosclerosis and chronic obstructive pulmonary disease. SCAPIS 2 will investigate 15,000 study participants approximately 8-10 years after the baseline examination SCAPIS 1.

The five overall objectives of SCAPIS 2 are:

1. To determine characteristics related to the natural progression of atherosclerosis over 8-10 years.
2. To evaluate characteristics related to pathological cardiovascular aging over 8-10 years.
3. To determine characteristics related to the natural progression of lung function over 8-10 years.
4. To determine risk factors associated with the progression of coronary atherosclerosis and the development of impaired lung function or structural changes of the lungs.
5. To compare outcome in individuals who are invited to SCAPIS 2 and those not invited.

SCAPIS 2 will recruit approximately 15,000 subjects randomly selected from the baseline examination (SCAPIS 1) study population approximately 8-10 years after their initial participation. During the SCAPIS 1 random samples of men and women aged 50-64 years were drawn from each recruitment area in the Swedish population registry until approximately 30 000 subjects were included. The final number was 30 154 subjects with an even sex and age distribution. The original recruitment process ensured that the study population in SCAPIS 1 was representative for the Swedish population in general.

An invitation letter with brief information about SCAPIS 2 will be sent to randomly selected individuals by mail, including phone number and e-mail address to the study center. The invitation letter will refer to a study webpage where the subjects can indicate if they are interested in participating in SCAPIS 2 and read the subject information in advance (voluntary). The invitation also includes contact information to the study center to be used if the subject prefers to not use the web page or has questions. Subjects that have moved since their participation in SCAPIS 1 will be invited to the same study center as their baseline examination.

The examinations will be performed during 2-3 days within approximately 2 weeks. Whenever possible, all visits should be performed within a period of 4 weeks. Examinations that are common for all sites include:

* Medical history
* Anthropometry
* Clinical chemistry/hematology: Hb, p-Glucose, HbA1c, s-TG, s- Cholesterol, LDL, HDL, creatinine, detailed leukocyte count)
* Biobank sampling (plasma, serum, whole blood, and urine)
* Spirometry
* CO uptake
* Questionnaires
* Accelerometry (hip)
* Electrocardiogram (ECG)
* Heart rate
* Blood pressure
* Computed tomography (CT)

  * Body composition
  * Lung tissue
  * Coronary artery calcium score (CACS)
  * Coronary computed tomography angiography (CCTA)

All subjects will be fasting overnight (at least 8 hours) before the first visit. If a subject has not been fasting overnight, blood sampling should be rescheduled and performed preferably at an extra visit but no later than Visit 2. For subjects with elevated plasma glucose levels, an overnight fasting glucose measurement will be repeated.

Subjects should be instructed to take their regular medication as usual also when fasting. The only medication that should not be taken is medication for diabetes, per oral as well as injections. Subjects with diabetes should be fasting as all other subjects and should bring their medication to take when having breakfast at the clinic. To obtain standardized conditions for the CT examination, subjects are recommended to be fasting for at least 4 hours before intake of a standardized meal. The standardized meal should be consumed 2 hours before the CT scan.

All clinical findings and assessment of risk should be taken care of according to current guidelines and SCAPIS manual.

ELIGIBILITY:
Inclusion Criteria:

- Participated in SCAPIS 1.

Exclusion Criteria:

* Individuals who have withdrawn their informed consent during or after SCAPIS 1.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In the Swedish CArdioPulmonary bioImage Study (SCAPIS 1), 30,154 randomly selected men and women, aged 50-64 years, were recruited from six areas in Sweden during 2013-2018. The study population was investigated with CCTA, ultrasound carotids, physical examination, questionnaires, accelerometry, ECG, spirometry, and biochemical markers. The aim was to obtain new information relevant to the identification and treatment of individuals with cardiopulmonary and metabolic diseases and to optimize the possibilities for studying disease mechanisms.
  In SCAPIS-2, half of the individuals (n≈15,000) included in SCAPIS 1, will be re-examined 2024-2025 with the same investigations as during 2013-2018 except for ultrasound of the carotids.
Sampling Method: Probability Sample
Enrollment: 30154 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular death, non-fatal myocardial infarction or stroke. | Through study completion, an average of 5 years
  Cardiovascular death, non-fatal myocardial infarction or stroke.

SECONDARY OUTCOMES:
Cardiovascular death or non-fatal myocardial infarction | Through study completion, an average of 5 years
  Cardiovascular death or non-fatal myocardial infarction
Cardiovascular death | Through study completion, an average of 5 years
  Cardiovascular death
Myocardial infarction (fatal or non-fatal) | Through study completion, an average of 5 years
  Myocardial infarction (fatal or non-fatal)
Stroke (fatal or non-fatal) | Through study completion, an average of 5 years
  Stroke (fatal or non-fatal)
Death (all-cause) | Through study completion, an average of 5 years
  Death (all-cause)
Unstable angina requiring revascularization | Through study completion, an average of 5 years
  Unstable angina requiring revascularization
Chronic obstructive pulmonary disease (COPD) | Through study completion, an average of 5 years
  Chronic obstructive pulmonary disease (COPD)
Lung cancer | Through study completion, an average of 5 years
  Lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Carl Johan Östgren, PhD, Principal Investigator — Linkoeping University
Locations (6):
- Sweden (6):
  - Gothenburg University, Gothenburg
  - Linköping University, Linköping
  - Lund University, Lund
  - Karolinska Institutet, Stockholm
  - Umeå Universitet, Umeå
  - Uppsala University, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data can be shared if approved the Swedish Ethical Review Authority and authority responsible for personal data
Supporting Information: Study Protocol, ICF
Time Frame: After study completion
Access Criteria: Approval from the Swedish Ethical Review Authority and authority responsible for personal data

REFERENCES:
- [Background] Bergstrom G, Berglund G, Blomberg A, Brandberg J, Engstrom G, Engvall J, Eriksson M, de Faire U, Flinck A, Hansson MG, Hedblad B, Hjelmgren O, Janson C, Jernberg T, Johnsson A, Johansson L, Lind L, Lofdahl CG, Melander O, Ostgren CJ, Persson A, Persson M, Sandstrom A, Schmidt C, Soderberg S, Sundstrom J, Toren K, Waldenstrom A, Wedel H, Vikgren J, Fagerberg B, Rosengren A. The Swedish CArdioPulmonary BioImage Study: objectives and design. J Intern Med. 2015 Dec;278(6):645-59. doi: 10.1111/joim.12384. Epub 2015 Jun 19. PMID 26096600
- See also: website — https://www.scapis.org/